CLINICAL TRIAL: NCT07385586
Title: In Vivo Study for the Evaluation of the Efficacy of an Adjunct Mouthwash in Hygiene, Wound Healing, Analgesia, and Functional Recovery Following Trauma or Dental Procedures in Gingival Tissue
Brief Title: Evaluation of Mouthwash Use in Hygiene and Recovery After Interventions in Gums
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lacer S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nº23-003-1
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Damaged Oral Mucosa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repairing mouthwash (Experimental): Repairing mouthwash was used 3 times a day during 15 days after the procedure
  Interventions: Other: Repairing mouthwash
- Placebo (Placebo Comparator): Placebo was used 3 times a day during 15 days after the procedure
  Interventions: Other: Placebo mouthwash

INTERVENTIONS:
Other: Repairing mouthwash — repairing mouthwash was used 3 times a day for 15 days after dental procedure
  Arms: Repairing mouthwash
Other: Placebo mouthwash — placebo mouthwash was used 3 times a day for 15 days after dental procedure
  Arms: Placebo

SUMMARY:
The goal of this study was to learn if mouthwash works in aiding the healing of the gum tissue after trauma or dental procedure. The main questions it aims to answer are:

* Does mouthwash aid the healing of gum tissue?
* Does mouthwash help to reduce the pain?
* Is the mouthwash well accepted by the volunteers? Researchers will compare mouthwash to a placebo (a look-alike substance that contains no active ingredient) to see if mouthwash works to improve gum tissue healing.

Participants will:

* Use mouthwash or a placebo every day for 15 days
* Visit the dental clinic once a week for evaluations
* Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA I and II),
* both sexes,
* over 18 years old
* undergoing oral surgery (extractions, implants, etc.)
* wish to participate in the study.

Exclusion Criteria:

* Patients undergoing healing with Platelet-Rich Plasma (PRP).
* Allergy or hypersensitivity to any of the product's components.
* Patients under psychiatric treatment.
* Pregnant or breastfeeding women.
* Treatment with NSAIDs, analgesics, or antibiotics for other conditions at the time of starting the study.
* Treatment with healing antiseptics or oral hygiene products for other oral problems.
* Treatment with oral anticoagulants.
* Diabetics.
* Periodontal disease or an active infectious or acute inflammatory local process at the time of starting the study.
* Active smoking of more than 10 cigarettes per day.
* Poor oral hygiene.
* Any other condition deemed relevant by the specialist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Healing evaluation | The parameters were evaluated after the procedure and after 7 and 15 days of product use.
  Healing of the oral mucosa after the dental procedure was evaluated by the dentist on a 3 grade Likert scale (0 was good, 1 was acceptable, 2 was bad) taking into account wound edges, oral mucose colour and wound closure. The reduction of the score corresponded to improvement if the wound healing.

SECONDARY OUTCOMES:
Pain intensity evaluation | Pain was evaluated y subjects on a daily basis from procedure until day 7.
  Pain was evaluated on a scale from 0 to 10, where 0 is no pain and 10 is the maximum pain. Reduction of the number corresponded to pain improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Gala Servicios Clínicos, S.L.U., Don Benito, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No
The results of the study will be shared in the publication.

DOCUMENTS (1):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT07385586/Prot_000.pdf